CLINICAL TRIAL: NCT02566629
Title: Microbiota Community of Irritable Bowel Syndrome in Episodes and Remission Phase
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Other Study IDs: 2015SDU-QILU-G11
Record Dates: First submitted 2015-09-30; First posted 2015-10-02 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Irritable Bowel Syndrome
Keywords: microbiota community; IBS
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — extract 16S rDNA from fecal microflora
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- IBS patients in episodes phase: collect faeces from IBS patients in episodes remission phase
  Interventions: Other: collect faeces from participants
- IBS patients in remission phase: collect faeces from IBS patients in remission phase
  Interventions: Other: collect faeces from participants
- healthy controls: collect faeces from healthy controls
  Interventions: Other: collect faeces from participants

INTERVENTIONS:
Other: collect faeces from participants — analyze the fecal microbiota community using 16S rDNA detection technique

SUMMARY:
Analyze microbiota community of irritable bowel syndrome in episodes phase and remission phase.

DETAILED DESCRIPTION:
The pathophysiology of IBS is incompletely understood, it may involve an altered intestinal microbiota. Since the microflora composition of IBS is various in different studies, The investigators plan to compare the intestinal microbiota of IBS patients in episodes phase and remission phase with healthy controls,trying to find the difference.

ELIGIBILITY:
Inclusion Criteria:

* the presence of Rome III criteria for IBS ;
* Patients scheduled for colonoscopy examination or having negative screening examinations
* Aged between 18 and 65 years old

Exclusion Criteria:

* Antibiotic, probiotic or laxative usage within 4 weeks.
* organic gastrointestinal diseases
* Severe systematic disease: diabetes mellitus, hepatic, renal or cardiac dysfunction, thyroid disease or tumor etc.
* pregnancy or lactation.
* previous major or complicated abdominal surgery.
* severe endometriosis and dementia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients who fulfil the Rome III criteria of irritable bowel syndrome in Qilu Hospital outpatient
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-07; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
microbiota community among IBS patients in episodes phase,remission phase and healthy controls | 5 months

SECONDARY OUTCOMES:
quality of life in IBS patients | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, MD.PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China